CLINICAL TRIAL: NCT02031523
Title: A Randomized, Double-blind, Placebo-controlled Post-marketing Study to Assess the Treatment Effect of Sanjie Analgesic Capsule in Treating Endometriosis - Associated Pain
Brief Title: Multi-center Clinical Trials of Sanjie Analgesic Capsule in Treating Endometriosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NO.2-20130301
Record Dates: First submitted 2013-12-16; First posted 2014-01-09 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2013-12

CONDITIONS: Dysmenorrhea
Keywords: endometriosis; dysmenorrhea; Sanjie analgesic capsule; effect/safety
MeSH Terms: conditions — Dysmenorrhea; Endometriosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sanjie analgesic capsule (Active Comparator): every 4 capsules , 3 times a day, on the first day of menstruation to start taking, taking three consecutive menstrual cycle.
  Interventions: Drug: Sanjie analgesic capsule
- placebo (Placebo Comparator): every 4 capsules, 3 times a day, on the first day of menstruation to start taking, taking three consecutive menstrual cycle.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sanjie analgesic capsule — Oral, four each time, 3 times a day, on the first day of menstruation to start taking, taking three consecutive menstrual cycle.or follow the doctor's advice.
  Other Names: Jiangsu Kanion Pharmaceutical Co.,Ltd
  Arms: Sanjie analgesic capsule
Drug: placebo — oral，four each time, 3 times a day, on the first day of menstruation to start taking, taking three consecutive menstrual cycle. Or Follow the doctor's advice.
  Other Names: Jiangsu Kanion Pharmaceutical Co.,Ltd
  Arms: placebo

SUMMARY:
It is a multi-center, double -blind, placebo -controlled, randomized post-marketing study in Chinese subjects with endometriosis-associated pain to assess treatment effect and safety in the subjects treated with Sanjie Analgesic Capsule versus subjects treated with placebo.

DETAILED DESCRIPTION:
Sanjie Analgesic Capsule is a Chinese Traditional Patent Medicine. It is a botanical extract from the raw materials of the Resina Draconis , Panax Notoginseng, fritillary bulb and coix seed, which are derived from a classic prescription of traditional Chinese medicine.

Sanjie Analgesic Capsule was approved by CFDA in 2004, produced by means of modern technology by Jiangsu Kanion Pharmaceutical Co., Ltd. The study is a multi-center, double -blind, placebo-controlled, randomized in Chinese subjects with endometriosis-associated pain to assess treatment effect and safety in the subjects treated with Sanjie Analgesic Capsule versus subjects treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have a diagnosis of endometriosis by laparoscopy within 5 years prior to signing ICF, main complain of dysmenorrhea (or menstrual pain or painful periods) and with VAS score of 4 or above; Endometriosis combined with uterine adenomyosis is included.
* Female between the ages of 18 and 45 years old;
* Regular menstrual period, menstrual cycle falls in the ranging from 28 to 30 days;
* No pregnancy planning during taking study medication; use (or have their partner use) an acceptable method of birth control within the projected duration of the study ;
* Subjects must sign ICF and agree for follow up.

Exclusion Criteria:

* Genital cancer or other malignant tumor;
* Adnexal masses≥5cm;
* Uterine myoma≥3cm;
* Suffering from cardiovascular, hepatic, renal or hematopoietic system disease or mental illness;
* Receiving hormone therapy within 3 months prior to signing ICF;
* Receiving surgical treatment for endometriosis within 3 months prior to signing ICF;
* Subjects have a plan of pregnancy, being pregnant, breast-feeding during recent 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
dysmenorrhea | Baseline, 1,2,3,4 menstrual cycle

SECONDARY OUTCOMES:
change of Symptom (CPP Dyspareunia Defecate-pain Anal-bulge ) | baseline，1,2,3,4 menstrual cycle
change of Signs(Pelvic-tenderness Tubercle ) | baseline，1,2,3,4 menstrual cycle
change of Menstrual cycle and quantity | baseline，1,2,3,4 menstrual cycle
change of serum CA125 | baseline,3,4 menstrual cycle
the size of uterus and endometriosis cyst | baseline,3,4 menstrual cycle
change of serum endocrinological hormone | baseline,3,4 menstrual cycle
  the content of FSH, LH, E2, PRL, P, T
change of SF-36 score | Baseline,3 menstrual cycle
Safety assessments will be based on electrocardiogram, physical examinations, and clinical laboratory tests | Baseline,3 menstrual cycle
Safety assessments will be based on adverse event reports | 1,2,3 menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Lang Jinghe, Doctor, Principal Investigator — Beijing Union Medical College Hospital, Chinese Academy of Medical Sciences
Locations (14):
- China (14):
  - Beijing ChaoYang Hospital, Beijing, Beijing Municipality
  - Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The General Hospital of People's Liberation Army, Beijing, Beijing Municipality
  - Hubei Provincal Hospital of TCM, Wuhan, Hubei
  - The First Hospital of Hunan University of chinese Medicine, Changsha, Hunan
  - The Maternal and Child Health Hospital of Hunan Province, Changsha, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Jinan municipal hospital of Traditional Chinese Medicine, Jinan, Shandong
  - The Second Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Guangxing Hospital Of Zhejiang Chinese Medicine University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Leng JH, Duan H, Guan Z, Zhou YF, Qu H, Xu KH, Zhang SF, Zhang Q, Wang X, Lin KQ, Lang JH. Efficacy and Safety of Sanjie Analgesic Capsule in Patients with Endometriosis-Associated Pain: A Multicenter, 3:1 Randomized, Double-Blind, Placebo-Controlled Trial. Chin J Integr Med. 2024 Sep;30(9):780-787. doi: 10.1007/s11655-024-3756-y. Epub 2024 Jul 24. PMID 39046647